CLINICAL TRIAL: NCT02601248
Title: Single Site, Open-label, Dose Escalation Phase I Study of Theliatinib (HMPL-309) in Patients With Advanced Solid Tumors
Brief Title: Study of Theliatinib (HMPL-309) in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-309-00CH1
Record Dates: First submitted 2013-10-14; First posted 2015-11-10 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Cancer
Keywords: safety, PK
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Theliatinib (Experimental): Theliatinib investigational product once a day (QD) will be orally administrated on a 28-day cycle There are 5 dose cohorts,including120mg/160mg/200mg/220mg/300mg, QD in the dose escalation stage .
  Interventions: Drug: Theliatinib

INTERVENTIONS:
Drug: Theliatinib — Theliatinib is a tablet in the form of 25 mg ,10mg and 100 mg,oral,once daily
  Other Names: HMPL-309

SUMMARY:
First-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity(DLT), safety and tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of Theliatinib .

DETAILED DESCRIPTION:
Theliatinib (HMPL-309) is a new constructive, high effective, high selective, EGFR tyrosine kinase inhibitor. Theliatinib has demonstrated strong inhibitory effects on multiple tumors with overexpressed EGFR or sensitive EGFR mutations. This first-in-human study is conducted to assess the maximum tolerated dose (MTD) and dose-limiting toxicity(DLT), safety and tolerability, pharmacokinetics (PK), and preliminary anti-tumor activity of Theliatinib .

ELIGIBILITY:
Inclusion Criteria:

* Histopathology confirmed solid tumors
* Failed to standard treatment or no standard treatments for uncontrolled, recurrent and/or metastatic advance tumor (whatever previous surgery conditions)
* Age 18-75
* Performance status of 0, or 1, and no worse within 7days
* Life expected >3 months
* Written informed consent form voluntarily

Exclusion Criteria:

* Lab testing within 1 week before enrolled, AND<1.5×109/L, platelet<75×109/L, or Hb<9g/dL,
* Total bilirubin≥1.5× the upper limit of normal,
* Serum creatinine higher than normal range
* Diastolic pressure≥150mmHg or systolic pressure≥100mmHg whatever anti-hypertension drug used,
* Serum potassium (whenever potassium implemented) , serum calcium(ionic or albumin-type calcium) or serum magnesium outside normal ranges(whenever implemented)
* Within previous 4 weeks treated by systemic anti-tumor therapy, or radiotherapy, immune therapy, biological or hormonal therapy, and clinical trials. But exclude the below therapy, Prostate cancer treated by hormonal therapy such as GnRH analogue or antagonist Hormone replacement therapy or oral contraceptive Palliative radiotherapy for bone metastasis within 2 weeks
* Prior documental evidence of resistance to(epidermal growth factor receptor-tyrosine kinase inhibitors)
* Unrecovered from any previous therapy related toxicity to≤ CTCAE(Common Toxicity Criteria for Adverse Effects) 0 or 1or unrecovered from any previous surgery
* Any CNS(central nervous system) metastasis with uncontrolled symptoms
* Known dysphagia or drug malabsorption
* Active infections such as acute pneumonia, hepatitis B active period
* APTT (activated partial thromboplastin time) and/or INR(international normalized ratio), PT≥2 ULN (the upper limit of normal)(not including patients treated by anticoagulation treatment)
* ocular surface diseases or dry eye syndrome
* skin disease with obvious symptoms and signs
* significant cardiovascular disease, including II-IV atrioventricular block, acute myocardial infarction within 6 months, significant angina or Coronary artery bypass graft
* Known existing interstitial lung disease
* Female patients who are pregnant or feeding, or childbearing potential patient with pregnant testing positive
* Any abnormal of clinical and laboratory so that patients unsuitable to attend the trial sine in the opinion of the investigator
* Patients unable to comply with the protocol since significant psychological or psychogenic abnormal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Safety :the incidence of all adverse events by type and grade, abnormal laboratory changes | from day 1 of first dosing to 30days after permanent discontinuation of Thialitinib
  for each patient, adverse events are collected from the date of consent until 30 days after trial discontinuation

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) | Day 1-3 Single Dose and Day 1-28 Steady State
  Based on single-dose PK result, multi-dose stage subjects take HMPL-309 once a day or twice a day, PK samples are collected of a single oral dose of HMPL-309 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 28-Day cycle of therapy
Peak Plasma Concentration (Cmax) | Day 1-3 Single Dose and Day 1-28 Steady State
  Based on single-dose PK result, multi-dose stage subjects take HMPL-309 once a day or twice a day, PK samples are collected of a single oral dose of HMPL-309 on Day 1 to Day 3. At multiple-dose, Pharmacokinetics(PK) sampling will include a pre-dose and at the 0.5,2,4,6,8 hour time points on days 1,15,21of dosing in the first 28-Day cycle of therapy, and pre-dose on days 2,8,16,and 22 of the first 28-Day cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Su, PhD, Study Chair — Hutchison Medipharm Limited
Locations (1):
- Tianjin Cancer Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No